CLINICAL TRIAL: NCT03765164
Title: Glucose Control Using 1,5-AG: Randomized Controlled Trial
Brief Title: Glucose Control Using 1,5-AG Testing
Acronym: GLUCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qure Healthcare, LLC (Industry)
Collaborators: GlycoMark, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00024791
Record Dates: First submitted 2018-11-30; First posted 2018-12-05 (Actual); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The study is a pre-post, two-round, randomized controlled study of a nationally representative sample of primary care physicians, including internists and family physicians, randomly assigned to a control or intervention arm. Once eligibility is determined and providers are enrolled in the study, they will be asked to complete a questionnaire describing their practice and professional background. They will then care for a total of 6 CPV® simulated patients over the two rounds (3 per round). The simulated patients are adults aged 18-75 who present with diabetes, different levels of glycemic control and various co-morbidities. The study design consists of two study arms, a control arm and an intervention-arm that receives educational materials and the 1,5-AG results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (Active Comparator): Control participants will care for the same set of CPV patients as the intervention arm, but will not have knowledge of or access to GlycoMark 1,5-AG test results. Investigators will compare control participants' clinical recommendations to those in the intervention arm.
  Interventions: Other: Clinical Performance and Value Vignettes
- Intervention (Experimental): Intervention participants will care for the same set of CPV patients as the control arm, but will be educated on and given access to GlycoMark 1,5-AG test results. Investigators will compare intervention participants' clinical recommendations to those in the control arm.
  Interventions: Diagnostic Test: GlycoMark 1-5-AG; Other: Clinical Performance and Value Vignettes

INTERVENTIONS:
Diagnostic Test: GlycoMark 1-5-AG — Online educational materials on GlycoMark 1,5-AG and sample test results for simulated patients
  Arms: Intervention
Other: Clinical Performance and Value Vignettes — Simulated diabetic patients cared for online
  Other Names: CPVs

SUMMARY:
Glycemic excursions (temporary increases in blood glucose) are associated with health complications. Standard tests for diabetes (e.g. random blood sugar and HbA1c) do not test for these excursions despite their association with several health complications. GlycoMark's 1,5-anhydroglucitol (1,5-AG) is a validated indicator of glucose excursions in addition to short-term (1-2 weeks) hyperglycemia.

This study is a pre-post, two-round randomized controlled study of a nationally representative sample of primary care physicians. Investigators will assess whether physician participants are able to identify and address glycemic variability and hyperglycemia in their patients and, when given access to GlycoMark assay results, improve their patient management decisions by taking steps to optimize glycemic control, and reduce unnecessary resource utilization.

DETAILED DESCRIPTION:
Nearly half of the adult population, 114 million Americans, are diagnosed with diabetes or pre-diabetes, making it one of the most important public and personal health problems. Diabetes is the 7th leading cause of death in America and a contributing factor in many more deaths and lost days of productivity. Its complications include vascular disease, cardiovascular disease, stroke and dementia. The cost of diabetes care and its complications lead to $176 billion in direct medical costs and $69 billion in reduced productivity. With an over 2-fold increase in diabetes prevalence in the past two decades and an estimated 1.5 million new cases expected annually, it is clinically and economically critical for this condition to be managed appropriately.

Diabetes treatment programs focus on controlling hyperglycemia (random glucose > 200 mg/dL) without causing hypoglycemia (glucose < 70 mg/dL). Glucose control is determined in a number of ways in current clinical practice. Immediate and fasting blood sugars are determined in routine chemistry tests. The standard measure of long-term diabetes control, HbA1c testing, provides a reliable reading of average blood glucose levels over a 2-3-month period. In patients with high HbA1c levels, HbA1c measurement guides management decisions and helps the clinician bring the long-term glucose levels under control in poorly controlled diabetic patients. Random blood sugars and HbA1c is limited in that they do not reflect glycemic control in intervals greater than the past few hours and 2-3 months. In particular, they do not provide an indication of frequent, temporary increases in blood glucose, termed glycemic excursions, which have been independently associated with several health complications. Since it takes months for HbA1c levels to stabilize, HbA1c levels are also not helpful for patients starting medication or changing drug therapy.

1,5-anhydroglucitol (1,5-AG) is a molecule found in the blood and is a validated indicator of glucose excursions and short-term (1-2 weeks) hyperglycemia. In healthy patients without diabetes, or those with well-controlled diabetes, 1,5-AG is maintained at a steady state in the blood. However, during glycemic excursions, the molecule is actively purged from the body through the urine. Cleared by the FDA in 2003, the GlycoMark assay measures 1,5-AG levels in the blood. Low levels of 1,5-AG indicate the presence of potentially harmful glycemic excursion over the last 1 to 2 weeks, which may have been missed during random blood glucose testing and not sensitively detected by HbA1c.

GlycoMark testing provides clinical details on peak glucose levels, daily spikes, and response to drugs, including short term effects, of hypoglycemic agents that are otherwise not available, giving physicians a more complete understanding of their patient's glycemic control. This information may be clinically useful to help physicians make better management decisions, improve diabetes outcomes, avoid complications and reduce unnecessary spending.

This study is a pre-post, two-round randomized controlled study of a nationally representative sample of primary care physicians randomly assigned to a control or intervention arm. Enrolled participants will be asked to care for a sample of CPV® simulated patients. The simulated patients are adults aged 18-75 who present with diabetes, different levels of glycemic control and various co-morbidities. Participants randomized into an intervention-arm will receive educational materials and 1,5-AG test results when caring for their patients in round 2. Investigators will assess the participants' ability to identify and address glycemic variability and hyperglycemia and evaluate whether physicians who have access to GlycoMark take steps to optimize glycemic control and reduce unnecessary resource utilization.

ELIGIBILITY:
Inclusion Criteria:

* A minimum of 2 years post residency but no more than 30 years in practice
* Board-certified in internal medicine or family practice, primary care physicians
* In a private solo or multi-group practice
* Minimum threshold of patients (40+) currently seen weekly
* A minimum of 15% of their panel under their care for diabetes
* Have not used GlycoMark assay in the past
* Informed, signed and voluntarily consented to be in the study

Exclusion Criteria:

* Not board certified in their respective area of care
* Academic-based practice
* Have practiced as a board-certified physician for less than 2 or greater than 30 years
* Have used the GlycoMark assay
* Follow <40 patients weekly
* < 15% of their patient panel under their care for diabetes
* Non-English speaking
* Unable to access the internet

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-02-24 (Actual); Study Completion 2019-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Tran, MS, Study Director — QURE Healthcare; John W Peabody, MD, Principal Investigator — QURE Healthcare
Locations (1):
- QURE Healthcare, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Pre-intervention
Arm/Group | Control | Intervention
Started | 78 | 78
Completed | 73 | 72
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 5 | 6
Period: Post-intervention
Arm/Group | Control | Intervention
Started | 73 | 72
Completed | 0 | 0
Not Completed | 73 | 72

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 73 | 72 | 145
Age, Customized [Count of Participants; unit: Participants]
  <40 | 5 | 3 | 8
  40-55 | 45 | 42 | 87
  >55 | 23 | 27 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 18 | 29
  Male | 62 | 54 | 116
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Practice locale (urban, suburban, or rural) [Count of Participants; unit: Participants]
  Urban | 14 | 24 | 38
  Suburban | 45 | 33 | 78
  Rural | 14 | 15 | 29
U.S. Region Location of Practice [Count of Participants; unit: Participants]
  Midwest | 20 | 13 | 33
  Northeast | 17 | 13 | 30
  South | 22 | 30 | 52
  West | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Diagnosis-Treatment
Description: Difference-in-differences regression analysis between the control and the intervention group's identification and treatment of hyperglycemia, as measured by the participants diagnostic and treatment CPV case domain scores. In each domain of a CPV (history, physical exam, workup, diagnosis and treatment), participants' care recommendations are evaluated against evidence-based care scoring criteria which can sum to a high potential score of up to 100% in each domain.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: CPV diagnosis-treatment percentage score
Arm/Group | Control | Intervention
Number analyzed (Participants) | 73 | 72
CPV diagnosis-treatment percentage score
  Round 2 | 31.7 (13.4) | 35.0 (15.0)
  Round 1 | 29.1 (12.3) | 31.9 (12.2)

2. Secondary Outcome: Quality of Care
Description: Difference-in-differences regression analysis between the control and the intervention group's overall quality of care scores. In each CPV case, participants' care recommendations are evaluated against evidence-based care scoring criteria which can sum to a high potential score of up to 100% in each case.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: CPV overall percentage score
Arm/Group | Control | Intervention
Number analyzed (Participants) | 73 | 72
CPV overall percentage score
  Round 2 | 51.4 (11.1) | 52.1 (12.3)
  Round 1 | 50.9 (10.0) | 48.9 (10.8)

3. Secondary Outcome: Workup Costs
Description: Difference-in-differences regression analysis between between the control and the intervention group in the average cost of diagnostic tests ordered.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: US$
Arm/Group | Control | Intervention
Number analyzed (Participants) | 73 | 72
US$
  Round 2 | 78 (156) | 37 (87)
  Round 1 | 54 (100) | 60 (116)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/72
Other Adverse Events (participants affected / at risk) | 0/73 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT03765164/Prot_SAP_000.pdf